CLINICAL TRIAL: NCT00529360
Title: Clofarabine in Combination With Cytarabine and Total Body Irradiation Followed by Allogeneic Stem Cell Transplantation in Children With Acute Lymphoblastic Leukemia and Acute Non-Lymphoblastic Leukemia
Brief Title: Allogeneic Stem Cell Transplant With Clofarabine, Ara-C and TBI for AML and ALL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L 9471
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia
Keywords: Acute Leukemia; Allogeneic Stem Cell Transplant; Clofarabine; Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): Part A will be the dose escalation phase to determine the MTD and/or safe/tolerated dose of clofarabine.
  Interventions: Drug: Clofarabine
- Part B (Experimental): Part B will accrue patients to further define the event free, disease free and overall survival at the MTD or safe/tolerated dose of clofarabine.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Dose escalation of clofarabine on Days -9, -8, -7, -6, -5: 1 - 30 mg/m2; 2 - 40 mg/m2; 2 - 46 mg/m2; 3 - 52 mg/m2
  Other Names: Clolar®
  Arms: Part A
Drug: Clofarabine — Use dose of clofarabine established in Part A to further define event free, disease free and overall survival.
  Other Names: Clolar®
  Arms: Part B

SUMMARY:
Hypothesis: Myeloablative conditioning using a dose escalation of clofarabine in combination with cytarabine (ARA-C) and total body irradiation (TBI) will lead to improved survival for previously untransplanted children and adolescents with acute lymphoblastic leukemia (ALL) and acute non-lymphoblastic leukemia (ANLL)followed by allogeneic stem cell transplantation (AlloSCT).

DETAILED DESCRIPTION:
Pediatric patients with ALL who have multiple relapses show a declining reinduction rate with each successive relapse. Chessels et al reported the results in 235 pediatric patients with ALL in CR3 treated between 1972 and 1998. Only 18 of the 235 patients remained alive, with multiple early treatment failures implying significant instability of the third remission state. Factors that were found to be of significant influence on survival for these patients in CR3 were length of CR2, type of second event, immunophenotype, type of third treatment, type of first relapse, presenting leukocyte count, and length of CR1. The 3-year leukemia-free survival for patients with ALL in CR3 treated with hematopoietic progenitor cell transplantation (HPCT) was reported as 20% in a single-institution report on patients transplanted with unrelated donors between 1987 and 1999. This report found a 20% relapse rate in ALL patients in CR3 and reported that patients transplanted after 1992 had a higher rate of relapse, implying that as improved chemotherapy regimens become more successful in curing patients, those who develop relapse may have disease more resistant to treatment. Clofarabine ([2-chloro-9-(2-deoxy-2-fluoro-D-arabinofuranosyl)adenine]; Cl-F-ara-A; CAFdA) is a rationally designed, second-generation purine nucleoside antimetabolite. Clofarabine was designed as a hybrid molecule to overcome the limitations and incorporate the best qualities of fludarabine (F-ara-A) and cladribine (2-CdA, CdA), all three molecules are currently approved by the FDA for treatment of hematologic malignancies. In an open-label Phase II, pediatric patients with refractory or relapsed ALL received clofarabine 52 mg/m2 by IVI over 2 hours for 5 consecutive days repeated every 2 to 6 weeks depending on toxicity and response. Among the 49 patients evaluated for efficacy, the overall remission rate was 20%. The median duration of remission could not be calculated for the 6 patients who achieved a CR because 3 patients were still in remission at the time of data cutoff. The median duration for the 4 patients who achieved a CRp was 20 weeks (Range: 4.6 to 28.6 weeks). Eight (16%) patients went on to receive a transplant with 7 (14%) experiencing clinical benefit. In an open-label Phase II study, pediatric patients with refractory or relapsed AML received clofarabine 52 mg/m2 by IVI over 2 hours for 5 consecutive days repeated every 2 to 6 weeks depending on toxicity and response. The overall remission rate (CR + CRp) was 3%; 23% of patients achieved a PR. The median duration of remission for patients who achieved at least a PR was 16.2 weeks. Twelve (34%) patients went on to receive a transplant, 7 of whom were still alive at the time of data cutoff with survival ranging from 16.4 weeks to 93.6 weeks.

Patients enrolling must have undergone an extensive pre-transplant evaluation to assess remission status, assure adequate organ system function, and document freedom from active viral, bacterial, and fungal infection. Patients should proceed to transplant as soon as possible following their reinduction chemotherapy. Patients with delays in therapy due to toxicity or donor procurement delays should receive maintenance chemotherapy if possible. Patients must be scheduled to begin their preparative regimen within 10 days of enrolling on the study. This will be a 2 part study. Part A will be the dose escalation phase. Once the MTD and/or safe/tolerated dose of clofarabine has been established, Part B will accrue patients to further define the event free, disease free and overall survival at the MTD or safe/tolerated dose of clofarabine. At study entry during Part A, a clofarabine dose level will be assigned to each patient. During Part B, the established MTD or safe/tolerated dose of clofarabine will be used.

In Part A this study will enroll patients with ALL and ANLL in relapse, induction failure, CR3 or CR3P and without prior AlloSCT. These patients will receive a conditioning regimen of clofarabine, ARA-C and TBI followed by AlloSCT. Patients will start their pre-conditioning regimen on Day -10. Patients will receive ARA-C (3000 mg/m2 [total ARA-C dose of 18g/m2]) daily on Days -10, -9, -8, -7, -6, and -5 and clofarabine (Dose assigned at enrollment, see section 8.2.2 for dose escalation table for Part A) on Days -9, -8, -7, -6, and -5. On days when clofarabine and ARA-C are both given, clofarabine will be given as a 2 hr infusion followed by 4 hr rest and then ARA-C given as a 3 hr infusion. Fractionated TBI (200 cGy) will be administered twice daily for 3 days on Day -4, -3 and -2. The AlloSCT will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus and MMF. In Part B, this study will enroll patients with ALL or ANLL in CR3 or CR3P and without prior AlloSCT. The pre-conditioning regimen will be the same as in Part A EXCEPT the established MTD or safe/tolerated dose of clofarabine from Part A will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be <30 years of age.
* Disease Status: ALL in relapse, induction failure, CR3, or CR3P (Part A ONLY); AML in relapse, induction failure, CR3, or CR3P (Part A ONLY); ALL in CR3 or CR3P (Part A and Part B); AML in CR3 or CR3P (Part A and BONLY); CR3/CR3P must be documented by bone marrow and CNS assessment within 14 days of initiation of the pre-transplant conditioning regimen.
* Creatinine clearance >40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent radioisotope glomerular filtration rate (GFR) as determined by the institutional normal range or serum creatinine based on age
* Adequate liver function defined as: Total bilirubin <2.5 mg/dl l, or SGOT (AST) or SGPT (ALT) <5 x upper limit of normal
* Adequate cardiac function defined as: Shortening fraction >27% by echocardiogram, or Ejection fraction of >50% by radionuclide angiogram or echocardiogram.
* Adequate pulmonary function defined as: Corrected DLCO >60% by pulmonary function test; For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air.
* Performance Status: For patients age 1-16 years, Lansky score of >60; For patients > 16 years, Karnofsky score of >60.
* Patients must have received a minimum of one round of re-induction and one round of consolidation chemotherapy after relapse #2

Exclusion Criteria:

* Patients with prior myeloablative allogeneic stem cell transplantation and /or TBI.
* Females who are pregnant (positive HCG) or lactating.
* Karnofsky <60% or Lansky <60% if less than 16 years of age
* Age >30 years of age
* Any patient with uncontrolled infection prior to study entry
* Patients with evidence of active disease.
* Patients with Down syndrome are excluded

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and/or the safe, tolerated dose of clofarabine in combination with ARA-C and TBI followed by AlloSCT in children with ALL and ANLL. | 2.5 years
To define the toxicity and safety of the conditioning regimen of clofarabine, ARA-C, TBI followed by AlloSCT in children with ALL and ANLL. | 2.5 years
To define the pharmacokinetics of clofarabine given in combination with ARA-C and TBI followed by AlloSCT in children with ALL and ANLL. | 2.5 years

SECONDARY OUTCOMES:
To determine the event-free, disease-free and overall survival of the conditioning regimen of clofarabine, ARA-C and TBI followed by AlloSCT in children with ALL and AML. | 5 years
To estimate the time to hematopoietic reconstitution, stratified by cell source, following clofarabine, ARA-C and TBI followed by AlloSCT in children with ALL and AML. | 2.5 years
To measure the changes in minimal residual disease with ALL and AML following clofarabine, ARA-C and TBI followed by AlloSCT | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Vallhala, New York, United States